CLINICAL TRIAL: NCT00636077
Title: Effect Of Dialysate Flow Rate On Mass Transfer Coefficient - Area (KoA) In Dialyzers With Different Membrane Packing Densities
Brief Title: Comparative Effects Of Dialysate Flow Rate And Membrane Packing On The Performance Of Dialyzers Used For Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: University of Louisville (Other); Gambro Renal Products, Inc. (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Gambro 1461
Record Dates: First submitted 2008-02-20; First posted 2008-03-14 (Estimated); Results first posted 2011-07-01 (Estimated); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Disease; Chronic Renal Disease
Keywords: Hemodialysis; Dialysis, Renal
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- HD-C4 Big (Other): 3 consecutive treatments with the HD-C4 Big dialyzer.
  Interventions: Device: Polyflux HD-C4 Big
- HD-C4 Small (Other): 3 consecutive treatments with the HD-C4 Small dialyzer.
  Interventions: Device: HD-C4 Small
- F160NR (Other): 3 consecutive treatments with the F160NR dialyzer.
  Interventions: Device: Optiflux 160NR
- F200NR (Other): 3 consecutive treatments with the F200NR dialyzer.
  Interventions: Device: Optiflux 200NR

INTERVENTIONS:
Device: Polyflux HD-C4 Big — Three consecutive treatments with the HD-C4 Big. During the third treatment, dialyzer clearances of urea, phosphorus and β2-microglobulin will be determined at a blood flow rate of 400 mL/min and dialysate flow rates of 350 mL/min, 500 mL/min and 800 mL/min.
  Other Names: Gambro Polyflux HD-C4 Big dialyzer; Gambro Revaclear MAX
  Arms: HD-C4 Big
Device: HD-C4 Small — Three consecutive treatments with the HD-C4 Small. During the third treatment dialyzer clearances of urea, phosphorus and β2-microglobulin will be determined at a blood flow rate of 400 mL/min and dialysate flow rates of 350 mL/min, 500 mL/min and 800 mL/min.
  Other Names: Gambro Polyflux HD-C4 Small dialyzer; Gambro Revaclear dialyzer
  Arms: HD-C4 Small
Device: Optiflux 160NR — Three consecutive treatments with the HD-C4 Small. During the third treatment dialyzer clearances of urea, phosphorus and β2-microglobulin will be determined at a blood flow rate of 400 mL/min and dialysate flow rates of 350 mL/min, 500 mL/min and 800 mL/min.
  Other Names: Fresenius Optiflux 160NR
  Arms: F160NR
Device: Optiflux 200NR — Three consecutive treatments with the HD-C4 Small. During the third treatment dialyzer clearances of urea, phosphorus and β2-microglobulin will be determined at a blood flow rate of 400 mL/min and dialysate flow rates of 350 mL/min, 500 mL/min and 800 mL/min.
  Other Names: Fresenius Optiflux 200NR
  Arms: F200NR

SUMMARY:
The purposes of this study are to determine if the performance of a dialyzer depends on how tightly the hollow fiber membranes are packed in the housing of the dialyzer (the membrane packing density) and if that dependence is a function of the dialysate flow rate. The study will examine how efficiently three different sized molecules pass through a dialyzer membrane at different dialysate flow rates in dialyzers with different membrane packing densities. Transfer of urea, phosphorus and beta-2-microglobulin from blood to dialysate will be measured during clinical hemodialysis using four different dialyzers, each used at three different dialysate flow rates. The data derived from these measurements may provide insight into the importance of membrane packing density as a design parameter for hemodialyzers and if changing the membrane packing density might provide equivalent performance at a lower dialysate flow rate.

ELIGIBILITY:
Inclusion Criteria:

* Stable hemodialysis patients dialyzing through a native fistula or Gore-Tex graft. The access must be capable of delivering a stable blood flow of 400 ml/min.
* Age older than 18 years.
* Fluid removal requirement less than 3 liters per treatment.

Exclusion Criteria:

* Noncompliance with dialysis regimen.
* Hematocrit less than 28%.
* Active infection

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-02; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Ward, Ph.D., Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Kidney Disease Program, Louisville, Kentucky, United States

REFERENCES:
- [Background] Leypoldt JK, Cheung AK, Agodoa LY, Daugirdas JT, Greene T, Keshaviah PR. Hemodialyzer mass transfer-area coefficients for urea increase at high dialysate flow rates. The Hemodialysis (HEMO) Study. Kidney Int. 1997 Jun;51(6):2013-7. doi: 10.1038/ki.1997.274. PMID 9186896
- [Background] Ouseph R, Ward RA. Increasing dialysate flow rate increases dialyzer urea mass transfer-area coefficients during clinical use. Am J Kidney Dis. 2001 Feb;37(2):316-20. doi: 10.1053/ajkd.2001.21296. PMID 11157372
- [Background] Michaels AS. Operating parameters and performance criteria for hemodialyzers and other membrane-separation devices. Trans Am Soc Artif Intern Organs. 1966;12:387-92. No abstract available. PMID 5960730
- [Background] Ward RA, Ouseph R: Comparative evaluation of small and large molecule removal during hemodialysis with Polyflux-S and Fresenius polysulfone membranes. Report to Gambro Renal Products, February 6, 2003.
- [Background] Ward RA, Ouseph R: A comparison of urea, phosphorus and b2-microglobulin removal during hemodialysis with dialyzers containing Polyflux H and Fresenius Optiflux membranes. Report to Gambro Renal Products, August 29, 2005.
- [Background] Leypoldt JK, Cheung AK, Chirananthavat T, Gilson JF, Kamerath CD, Deeter RB. Hollow fiber shape alters solute clearances in high flux hemodialyzers. ASAIO J. 2003 Jan-Feb;49(1):81-7. doi: 10.1097/00002480-200301000-00013. PMID 12558312
- [Background] Ward RA, Ouseph R: Modification of membrane characteristics allows a reduction in dialyzer membrane area without loss of performance. J Am Soc Nephrol 18:453A, 2007.
- [Background] Chen PS, Toribara TY, Warner H. Microdetermination of phosphorus. Anal Chem 1956; 28: 1756-1758
- [Result] Bhimani JP, Ouseph R, Ward RA. Effect of increasing dialysate flow rate on diffusive mass transfer of urea, phosphate and beta2-microglobulin during clinical haemodialysis. Nephrol Dial Transplant. 2010 Dec;25(12):3990-5. doi: 10.1093/ndt/gfq326. Epub 2010 Jun 13. PMID 20543211

RESULTS

PARTICIPANT FLOW:
Groups:
- HD-C4 Big First: Patients in this Arm will receive 3 consecutive treatments with the HD-C4 Big dialyzer first. For the study each patient will be treated for three consecutive treatments with each of the 4 study dialyzers (total of 12 consecutive treatments).
- HD-C4 Small First: Patients in this Arm will receive 3 consecutive treatments with the HD-C4 Small dialyzer first. For the study each patient will be treated for three consecutive treatments with each of the 4 study dialyzers (total of 12 consecutive treatments).
- Optiflux F160NR First: Patients in this Arm will receive 3 consecutive treatments with the F160NR dialyzer first. For the study each patient will be treated for three consecutive treatments with each of the 4 study dialyzers (total of 12 consecutive treatments).
- Optiflux F200NR First: Patients in this Arm will receive 3 consecutive treatments with the F200NR dialyzer first. For the study each patient will be treated for three consecutive treatments with each of the 4 study dialyzers (total of 12 consecutive treatments).
Period: Week 1
Arm/Group | HD-C4 Big First | HD-C4 Small First | Optiflux F160NR First | Optiflux F200NR First
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Week 2
Arm/Group | HD-C4 Big First | HD-C4 Small First | Optiflux F160NR First | Optiflux F200NR First
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Week 3
Arm/Group | HD-C4 Big First | HD-C4 Small First | Optiflux F160NR First | Optiflux F200NR First
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Week 4
Arm/Group | HD-C4 Big First | HD-C4 Small First | Optiflux F160NR First | Optiflux F200NR First
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: Years] | 60 [32 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Effect of Increased Dialysate Flow Rate on KoA for Urea Between 4 Dialyzers With Different Membrane Packing Densities.
Description: KoA is a constant that describes the efficiency of a dialyzer in removing urea. KoA is determined by surface area of the membrane, the thickness of the membrane and pore size.
Time Frame: During the third treatment with each dialyzer (one time during each trial period week)
Measure: Mean (Standard Error); unit: KoA for urea (mL/min)
Arm/Group | HD-C4 Big | HD-C4 Small | F160NR | F200NR
Number analyzed (Participants) | 12 | 12 | 12 | 12
KoA for urea (mL/min)
  350 mL/min Dialysate Flow Rate | 844 (30) | 763 (34) | 770 (36) | 798 (21)
  500 mL/min Dialysate Flow Rate | 898 (31) | 748 (34) | 738 (40) | 890 (33)
  800 mL/min Dialysate Flow Rate | 922 (31) | 761 (25) | 809 (24) | 817 (36)

2. Primary Outcome: Effect of Increased Dialysate Flow Rate on Whole Blood Urea Clearance Between 4 Dialyzers With Different Membrane Packing Densities.
Time Frame: During the third treatment with each dialyzer (one time during each trial period week)
Measure: Mean (Standard Error); unit: Whole blood urea clearance (mL/min)
Arm/Group | HD-C4 Big | HD-C4 Small | F160NR | F200NR
Number analyzed (Participants) | 12 | 12 | 12 | 12
Whole blood urea clearance (mL/min)
  350 mL/min Dialysate Flow Rate | 279 (3) | 270 (4) | 271 (4) | 274 (2)
  500 mL/min Dialysate Flow Rate | 315 (3) | 295 (5) | 293 (8) | 313 (4)
  800 mL/min Dialysate Flow Rate | 340 (3) | 320 (3) | 313 (4) | 327 (5)

3. Primary Outcome: Effect of Increased Dialysate Flow Rate on KoA for Phosphorus Between 4 Dialyzers With Different Membrane Packing Densities.
Time Frame: During the third treatment with each dialyzer (one time during each trial period week)
Measure: Mean (Standard Error); unit: KoA for Phosphorus (mL/min)
Arm/Group | HD-C4 Big | HD-C4 Small | F160NR | F200NR
Number analyzed (Participants) | 12 | 12 | 12 | 12
KoA for Phosphorus (mL/min)
  350 mL/min Dialysate Flow Rate | 434 (48) | 334 (24) | 434 (34) | 504 (58)
  500 mL/min Dialysate Flow Rate | 435 (31) | 422 (48) | 450 (62) | 491 (29)
  800 mL/min Dialysate Flow Rate | 520 (39) | 415 (35) | 458 (33) | 560 (40)

4. Primary Outcome: Effect of Increased Dialysate Flow Rate on Whole Blood Phosphorus Clearance Between 4 Dialyzers With Different Membrane Packing Densities.
Time Frame: During the third treatment with each dialyzer (one time during each trial period week)
Measure: Mean (Standard Error); unit: whole blood phosphorus clearance mL/min
Arm/Group | HD-C4 Big | HD-C4 Small | F160NR | F200NR
Number analyzed (Participants) | 12 | 12 | 12 | 12
whole blood phosphorus clearance mL/min
  350 mL/min Dialysate Flow Rate | 255 (7) | 252 (9) | 247 (6) | 249 (5)
  500 mL/min Dialysate Flow Rate | 269 (10) | 261 (9) | 260 (7) | 265 (7)
  800 mL/min Dialysate Flow Rate | 286 (7) | 273 (7) | 272 (7) | 281 (7)

5. Primary Outcome: Effect of Increased Dialysate Flow Rate on KoA for b2-microglobulin Between 4 Dialyzers With Different Membrane Packing Densities.
Time Frame: During the third treatment with each dialyzer (one time during each trial period week)
Measure: Mean (Standard Error); unit: KoA for b2-microglobulin (mL/min)
Arm/Group | HD-C4 Big | HD-C4 Small | F160NR | F200NR
Number analyzed (Participants) | 12 | 12 | 12 | 12
KoA for b2-microglobulin (mL/min)
  350 mL/min Dialysate Flow Rate | 65 (4) | 61 (2) | 27 (2) | 27 (2)
  500 mL/min Dialysate Flow Rate | 62 (3) | 57 (2) | 28 (2) | 25 (2)
  800 mL/min Dialysate Flow Rate | 64 (3) | 56 (3) | 31 (5) | 21 (1)

6. Primary Outcome: Effect of Increased Dialysate Flow Rate on Whole Blood B2-microglobulin Clearance Between 4 Dialyzers With Different Membrane Packing Densities.
Time Frame: During the third treatment with each dialyzer (one time during each trial period week)
Measure: Mean (Standard Error); unit: whole blood clearance B2-microglobulin
Arm/Group | HD-C4 Big | HD-C4 Small | F160NR | F200NR
Number analyzed (Participants) | 12 | 12 | 12 | 12
whole blood clearance B2-microglobulin
  350 mL/min Dialysate Flow Rate | 106 (9) | 119 (6) | 87 (6) | 72 (9)
  500 mL/min Dialysate Flow Rate | 129 (7) | 118 (8) | 86 (10) | 65 (5)
  800 mL/min Dialysate Flow Rate | 118 (7) | 121 (9) | 78 (8) | 75 (7)

ADVERSE EVENTS:
Arm/Group | HD-C4 Big | HD-C4 Small | F160NR | F200NR
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No